CLINICAL TRIAL: NCT01707004
Title: Decitabine Followed by Bone Marrow Transplant and High-Dose Cyclophosphamide for the Treatment of Relapsed and Refractory Acute Myeloid Neoplasms
Brief Title: Decitabine and Total-Body Irradiation Followed By Donor Bone Marrow Transplant and Cyclophosphamide in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO11421; NCI-2012-01325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0217; 2017-0116; P30CA014520 (NIH); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison)
Record Dates: First submitted 2012-10-08; First posted 2012-10-15 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-05

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Decitabine; Azacitidine; fludarabine phosphate; Busulfan; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Filgrastim; Granulocyte Colony-Stimulating Factor; Whole-Body Irradiation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (donor bone marrow transplant) (Experimental): Beginning between days -29 and -22, patients receive decitabine IV over 1 hour daily for 10 days, fludarabine phosphate IV over 30 minutes on days -5 to -2, and busulfan IV over 3 hours on days -5 to -2.
  PREPARATIVE REGIMEN: Patients undergo total-body irradiation BID on day -1.
  TRANSPLANT: Patients undergo allogeneic bone marrow transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 2 hours on days 3 and 4, tacrolimus PO BID or IV continuously on days 5-180, mycophenolate mofetil PO TID on days 5-35, and filgrastim SC beginning day 5 until ANC >= 1,000/mm^3 for 3 consecutive days.
  Interventions: Drug: decitabine; Drug: fludarabine phosphate; Drug: busulfan; Drug: cyclophosphamide; Drug: tacrolimus; Drug: mycophenolate mofetil; Biological: filgrastim; Radiation: total-body irradiation; Procedure: allogeneic bone marrow transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-2'-deoxycytidine (5-aza-dCyd); 5-azacytidine (5AZA); decitabine (DAC)
Drug: fludarabine phosphate — Given IV
  Other Names: Fludarabine phosphate (2-F-ara-AMP); Beneflur; Fludara
Drug: busulfan — Given IV
  Other Names: busulfan (BSF); busulfan (BU); Misulfan; Mitosan; Myeloleukon
Drug: cyclophosphamide — Given IV
  Other Names: cyclophosphamide (CPM); cyclophosphamide (CTX); Cytoxan; Endoxan; Endoxana
Drug: tacrolimus — Given PO or IV
  Other Names: tacrolimus (FK 506); Prograf
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; mycophenolate mofetil (MMF)
Biological: filgrastim — Given SC
  Other Names: granulocyte-colony stimulating factor (G-CSF); Neupogen
Radiation: total-body irradiation — Undergo total-body irradiation
  Other Names: total body irradiation (TBI)
Procedure: allogeneic bone marrow transplantation — Undergo allogeneic bone marrow transplantation
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well decitabine and total-body irradiation followed by donor bone marrow transplant and cyclophosphamide works in treating patients with relapsed or refractory acute myeloid leukemia. Giving decitabine and total-body irradiation before a donor bone marrow transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving decitabine and total-body irradiation before the transplant together with high-dose cyclophosphamide, tacrolimus, and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine overall survival at 100 days after transplantation following decitabine and a bone marrow transplant using a donor that is at least partially-matched and a myeloablative preparative regimen with post-transplantation cyclophosphamide for graft-versus-host disease (GVHD) prophylaxis.

SECONDARY OBJECTIVES:

I. Patients enrolled in this study will also be followed for the following endpoints: neutrophil and platelet recovery, graft failure, acute graft-versus-host disease (GVHD), chronic GVHD, incidence of infection, treatment-related mortality, time to relapse/progression, overall survival, and progression-free survival.

OUTLINE:

Beginning between days -29 and -22, patients receive decitabine intravenously (IV) over 1 hour daily for 10 days, fludarabine phosphate IV over 30 minutes on days -5 to -2, and busulfan IV over 3 hours on days -5 to -2.

PREPARATIVE REGIMEN: Patients undergo total-body irradiation twice daily (BID) on day -1.

TRANSPLANT: Patients undergo allogeneic bone marrow transplant on day 0.

GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 2 hours on days 3 and 4, tacrolimus orally (PO) BID or IV continuously on days 5-180, mycophenolate mofetil PO three times daily (TID) on days 5-35 and filgrastim subcutaneously (SC) beginning day 5 until absolute neutrophil count (ANC) >= 1,000/mm^3 for 3 consecutive days.

After completion of study treatment, patients are followed up at 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet one of two disease criteria:

  * Acute myelogenous leukemia (AML) within one of the following categories:

    * Primary induction failure (PIF): patients who have not achieved a complete remission following initial diagnosis and after at least two induction cycles of chemotherapy consisting of cytarabine and an anthracycline or high-dose cytarabine
    * Relapsed AML: Patients are defined as having relapsed disease if they entered a complete remission confirmed with a bone marrow biopsy following initial treatment, and then were found to have morphological or cytogenetic evidence of recurrent disease on a subsequent bone marrow exam
    * Any complete remission (CR) 2 or greater: CR must be defined using a bone marrow exam taken at least 21 days since the last chemotherapy (including a methyltransferase inhibitor), and may include CRp (morphologic CR without peripheral platelet recovery)
    * CR1 with high-risk features: includes patients with treatment-related AML, secondary AML (following myelodysplastic syndrome (MDS) or myeloproliferative neoplasms (MPN)), high-risk cytogenetic or molecular phenotype (by National Comprehensive Cancer Network (NCCN) criteria)
    * Untreated AML (> 20% blasts on a bone marrow) arising from a previous confirmed diagnosis of MDS or MPN (excluding BCR-ABL (a genetic mutation) positive diseases).
  * Myelodysplastic syndromes within one of the following categories:

    * High-risk myelodysplastic syndrome (MDS) at diagnosis as defined by the International Prognostic Scoring System (IPSS) or World Health Organization (WHO) classification based Prognostic Scoring System (WPSS)
    * Transfusion dependent MDS (either red blood cells (RBC) or platelet dependent) without a hematologic response to at least 4 months of methyltransferase inhibitor (MTI) therapy; hematological response is defined as transfusion independence for two or more months
    * Progressive MDS following at least 4 months of MTI therapy; progression is defined as resumption of transfusion dependence after at least two months of transfusion independence OR increase of marrow blasts by 50% from pretreatment OR overall blasts over 10% of marrow cells at any time after treatment
* Available related donor that is at least an allele level haplotype-match at human leukocyte antigen (HLA)- A, B, C, DP Beta 1 (DRB1) and DPB1 loci (DPB1 matching according to the "permissive - non-permissive" dichotomy as stated by University of Wisconsin (UW) Histocompatibility Laboratory); a minimum match of 5/10 loci is required; an unrelated donor search is not required for a patient to be eligible for this protocol
* Karnofsky score of 60% or better (requires occasional assistance, but is able to care for most of his/her needs)
* Diffusing capacity of the lungs for carbon monoxide (DLCO) (corrected for hemoglobin > 40%; and forced expiratory volume in one second (FEV1) > 50%
* Ejection fraction (EF) >= 50% and no uncontrolled angina, symptomatic ventricular arrhythmias, or electrocardiogram (ECG) evidence of active ischemia
* Serum creatinine within normal range for age, or if serum creatinine outside normal range, then renal function (estimated glomerular filtration rate (GFR) by modification of diet in renal disease (MDRD) formula) > 40 mL/min/1.73 m^2
* Women of child bearing potential must have a negative pregnancy test within 14 days prior to study registration and agree to use adequate birth control during study treatment
* Voluntary written consent
* Patients must be 28 days from the end of the last induction course or at least 14 days from completion of previous methyltransferase inhibitor therapy (azacitidine or decitabine) at the time of registration
* DONOR: Donors must be at least HLA-haploidentical first degree relatives of the patients; eligible donors include biological parents, siblings, half-siblings or children
* DONOR: Age >= 18 years and =< 60 years
* DONOR: Donors must meet the selection criteria prior to the start of the recipient's pre-transplant conditioning regimen as defined by the Foundation for the Accreditation of Cell Therapy (FACT) and will be screened according to the American Association of Blood Banks (AABB) guidelines and UW Bone Marrow Transplant (BMT) program standard operating procedure (SOP)

Exclusion Criteria:

* Active central nervous system (CNS) leukemia within two weeks of registration; patients with a history of CNS leukemia must have adequate treatment as defined by at least two negative spinal fluid assessments separated by at least one week; patients who have received cranial radiation therapy (XRT) must still be eligible to receive total body irradiation to 4 Gy
* New or active infection as determined by fever, unexplained pulmonary infiltrate or sinusitis on radiographic assessment; infections diagnosed within 4 weeks of registration must be determined to be controlled or resolving prior to treatment
* Active human immunodeficiency virus (HIV), hepatitis A, B or C infection
* Allergy or hypersensitivity to agents used within the treatment protocol
* DONOR: Recipient derived anti-donor high-titer (> 3000 MFI) HLA antibody as determined by Luminex assay
* DONOR: Not suitable for donation according to UW BMT program donor selection SOP

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2017-07-22 (Actual); Study Completion 2017-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Juckett, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Derived] D'Angelo CR, Hall A, Woo KM, Kim K, Longo W, Hematti P, Callander N, Kenkre VP, Mattison R, Juckett M. Decitabine induction with myeloablative conditioning and allogeneic hematopoietic stem cell transplantation in high-risk patients with myeloid malignancies is associated with a high rate of infectious complications. Leuk Res. 2020 Sep;96:106419. doi: 10.1016/j.leukres.2020.106419. Epub 2020 Jul 8. PMID 32683127
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of high risk BMT patients with active disease at time of transplant or very high risk to relapse post-transplant.
Groups:
- Decitabine + Bone Marrow Transplant: Pre-transplant Decitabine followed by Bone Marrow Transplant.
Period: Overall Study
Arm/Group | Decitabine + Bone Marrow Transplant
Started | 20
Completed | 17 (3 participants were not eligible to proceed to Bone Marrow Transplant due to significant infections.)
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine + Bone Marrow Transplant
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Donor Type [Count of Participants; unit: Participants] — Population: 17 participants received transplant on study
  Participants
    number analyzed (Participants) | 17
    Matched Related | 5
    Haplo-identical | 12
Disease Risk by DRI [Count of Participants; unit: Participants] — Disease Risk Index (DRI)
  Participants
    Low Risk | 0
    Intermediate Risk | 2
    High Risk | 13
    Very High Risk | 5
HCT-CI Score [Count of Participants; unit: Participants] — Hematopoietic Cell Transplantation Comorbidity Index (HCT-CI) - measures 17 categories of organ dysfunction. Total possible range is 0-29, the higher the number, the more co-morbidities. Higher comorbidity scores are associated with increased risk of transplant-related mortality.
  Participants
    0 | 5
    1-2 | 7
    3+ | 8
Disease Status [Number; unit: participants]
  AML | 15
  Primary Induction Failure | 6
  Relapsed Disease | 7
  CR1 with high risk features | 2
  MDS | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Will be analyzed using Kaplan-Meier (KM) method, and OS will be obtained from the KM estimates along with 95% confidence intervals.
Time Frame: Day 100
Population: (2 patients did not receive a transplant due to infectious complications, 1 patient received transplant off protocol)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Decitabine + Bone Marrow Transplant
Number analyzed (Participants) | 17
percentage of participants | 64.7 [45.5 to 91.9]

2. Secondary Outcome: Time to Neutrophil Recovery
Description: Defined as achieving an absolute neutrophil count (ANC) greater than or equal to 500/ul for three consecutive measurements on different days. Will be summarized with mean and standard deviation or median and interquartile range, and the change will be tested using a one-sample paired t-test at a two-tailed significance level of 0.05.
Time Frame: Up to 1 year
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Decitabine + Bone Marrow Transplant
Number analyzed (Participants) | 17
days | 16 [16 to 19]

3. Secondary Outcome: Percentage of Participants With Platelet Recovery by Day 30
Description: Platelet recovery is defined as the first day of a platelet count greater than 20,000/mm^3 with no platelet transfusions. Will be summarized with mean and standard deviation or median and interquartile range, and the change will be tested using a one-sample paired t-test at a two-tailed significance level of 0.05.
Time Frame: Up to day 30
Measure: Number (95% Confidence Interval); unit: percentage with plt engraftment, day 30
Arm/Group | Decitabine + Bone Marrow Transplant
Number analyzed (Participants) | 17
percentage with plt engraftment, day 30 | 58 [31.3 to 78.4]

4. Secondary Outcome: Number of Participants With Primary Graft Failure
Description: Defined as less than 5% donor chimerism in the cluster of differentiation (CD)3 and CD33 selected cell populations at any time after transplantation. Will be analyzed using KM method.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine + Bone Marrow Transplant
Number analyzed (Participants) | 17
Participants | 0

5. Secondary Outcome: Cumulative Incidence of Grade III-IV Acute GVHD
Description: Determined by the standard bone marrow transplant (BMT) Clinical Trials Network criteria (BMTCTN). Will be analyzed using KM method, a Graft versus Host Disease (GVHD) grade III-IV will be obtained from the KM estimates along with 95% confidence intervals.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Decitabine + Bone Marrow Transplant
Number analyzed (Participants) | 17
percentage of participants | 27.8 [8.0 to 52.3]

6. Secondary Outcome: Cumulative Incidence of Chronic GVHD According to BMTCTN
Description: Will be summarized with a proportion and a 95% confidence interval.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Decitabine + Bone Marrow Transplant
Number analyzed (Participants) | 17
percentage | 40.7 [6.9 to 74.0]

7. Secondary Outcome: Number of Participants With Complete Remission After Transplantation
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine + Bone Marrow Transplant
Number analyzed (Participants) | 17
Participants | 14

8. Secondary Outcome: Progression Free Survival
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Decitabine + Bone Marrow Transplant
Number analyzed (Participants) | 17
days | 141 [69 to 492]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) data were collected from registration to 1 year post-transplant.
Description: AEs were assessed at regularly scheduled follow up visits where physical exams and labs were performed. AEs reported here include grade 3-5 and adverse events that were not related to the disease state. AEs are reported for all participants who received Decitabine, 17 (+ 1 off protocol) participants who received the transplant.
Groups:
- Decitabine (N=20): Pre-transplant Decitabine
- Transplant (N=17): Pre-transplant Decitabine followed by Bone Marrow Transplant
Arm/Group | Decitabine (N=20) | Transplant (N=17)
All-Cause Mortality (participants affected / at risk) | 15/20 | 13/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 12/17
Other Adverse Events (participants affected / at risk) | 20/20 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (N=20) (N=20) | Transplant (N=17) (N=17)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 1
Encephalitis infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=20) (N=20) | Transplant (N=17) (N=17)
Anemia (Blood and lymphatic system disorders) | 20 (65) | 17 (202)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 6 (7)
Platelet Count Decreased (Investigations) | 18 (57) | 17 (139)
White Blood Cell Decreased (Investigations) | 17 (30) | 17 (105)
Neutrophil Count Decreased (Investigations) | 13 (30) | 17 (89)
Lymphocyte count decreased (Investigations) | 16 (30) | 16 (141)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 15 (31)
Alanine aminotransferase increased (Investigations) | 2 (2) | 12 (29)
Alkaline phosphatase increased (Investigations) | 5 (5) | 11 (22)
Creatinine increased (Investigations) | 3 (3) | 12 (26)
Weight loss (Investigations) | 2 (4) | 11 (42)
GGT increased (Investigations) | 1 (1) | 12 (26)
Blood bilirubin increased (Investigations) | 1 (1) | 10 (19)
Weight gain (Investigations) | 1 (1) | 6 (12)
INR increased (Investigations) | 0 (0) | 5 (6)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 2 (3)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 17 (37)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6) | 17 (80)
Hypokalemia (Metabolism and nutrition disorders) | 6 (12) | 16 (76)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5) | 17 (135)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 12 (28)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 11 (37)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 12 (25)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 9 (22)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 7 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 7 (11)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 8 (13)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 6 (15)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 7 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 11 (13) | 13 (39)
Edema limbs (General disorders) | 2 (2) | 13 (28)
Chills (General disorders) | 2 (2) | 7 (11)
Fever (General disorders) | 2 (2) | 3 (5)
Pain (General disorders) | 1 (1) | 3 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (4)
Facial pain (General disorders) | 1 (1) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 3 (3)
Localized edema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (12) | 15 (39)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 17 (49)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 15 (103)
Vomiting (Gastrointestinal disorders) | 2 (2) | 13 (43)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 11 (22)
Constipation (Gastrointestinal disorders) | 2 (2) | 10 (16)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 5 (5)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 4 (6)
Bloating (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (9)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 10 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (10)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (9)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 4 (4) | 12 (20)
Lung infection (Infections and infestations) | 3 (5) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (6)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (2)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (15) | 12 (88)
Hypotension (Vascular disorders) | 4 (4) | 9 (20)
Flushing (Vascular disorders) | 0 (0) | 2 (4)
Hematoma (Vascular disorders) | 1 (1) | 2 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 11 (11)
Dizziness (Nervous system disorders) | 2 (3) | 8 (14)
Headache (Nervous system disorders) | 3 (4) | 6 (10)
Tremor (Nervous system disorders) | 0 (0) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 5 (10)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (7)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (6)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 3 (3)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (3)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 6 (8) | 11 (30)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 6 (11)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 2 (4)
Delirium (Psychiatric disorders) | 0 (0) | 1 (3)
Dry eye (Eye disorders) | 0 (0) | 4 (5)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 3 (3)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 6 (11)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT01707004/Prot_SAP_000.pdf